CLINICAL TRIAL: NCT03479827
Title: Measuring the Peripheral Optical Quality of The Eye
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Geunyoung Yoon, Professor, University of Rochester
Other Study IDs: 71201
Record Dates: First submitted 2018-02-27; First posted 2018-03-27 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Nearsightedness
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Experimental: Subjects will undergo three Wavefront measurements, once with no contact lens, once with a monofocal contact lens and once with a bifocal contact lens.
  Interventions: Device: Monofocal Contact Lens; Device: Bifocal Contact Lens

INTERVENTIONS:
Device: Monofocal Contact Lens — A monofocal contact lens will be used for this measurement.
Device: Bifocal Contact Lens — A bifocal contact lens will be used for this measurement.

SUMMARY:
The goal of the study is to quantify wavefront aberration profiles of the eye with and without contact lens across the visual field. This will enable us to investigate the impact of the aberration on retinal image quality.

DETAILED DESCRIPTION:
The goal of this study is to investigate the effects of monofocal and bifocal soft contact lenses in the changes of peripheral optical quality and through-focus visual performance on real eyes. The goal will be accomplished by performing optical measurements using Shack-Hartmann wavefront sensor with and without the use of single vision and bifocal soft contact lenses.

ELIGIBILITY:
Inclusion Criteria

A person will be included in the study if he/she:

* Is 18 years or older and has full legal capacity to volunteer.
* Has no ocular condition or pathology, which may impact visual acuity e.g. keratoconus, amblyopia, cataract, macular degeneration;
* Has no active ocular disease or allergic conjunctivitis;
* Is not using any topical ocular medications;
* Is willing and able to follow instructions;
* Has voluntarily agreed to participate in the study by signing the statement of informed consent.

Exclusion Criteria

A person will be excluded from the study if he/she:

* Is under the age of 18 or over the age of 60 yrs.
* Correctable with high contrast logMAR acuity (EDTRS) testing to 20/20 or better;
* Pregnant at the time of enrolment in the study;
* Unable to handle, insert, remove or care for the study lenses;
* Considered by the Investigator to not be a suitable candidate for participation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults with no ocular pathology and uses contact lenses.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2020-11-29 (Actual); Study Completion 2020-11-29 (Actual)

PRIMARY OUTCOMES:
Mean Wavefront aberrations | less than 2 hours
  The scanning wavefront sensor will be used to collect data. Mean Wavefront aberrations for each trail will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Geunyoung Yoon, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No